CLINICAL TRIAL: NCT03952663
Title: Evaluation of the Effect of Platelet Rich Fibrin Membrane on the Neurosensory Dysfunction Following Inferior Alveolar Nerve Lateralization for Implant Placement"A Randomized Controlled Trial"
Brief Title: Effect of Platelet Rich Fibrin Membrane on the Neurosensory Dysfunction After IAN Lateralization for Implant Placement.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Sayed Ahmed Shalaby, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422015598557
Record Dates: First submitted 2019-05-07; First posted 2019-05-16 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Neurosensory Disorder
Keywords: inferior alveolar nerve lateralization; platelet rich fibrin; posterior atrophic mandible
MeSH Terms: conditions — Sensation Disorders

STUDY DESIGN:
Intervention Model Description: * Randomized clinical trial.
  * double blinded, with 1:1 allocation ratio, parallel design.
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded ,participant and outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): inferior alveolar nerve lateralization for dental implant placement ,and platelet rich fibrin membrane is placed around the nerve.
  Interventions: Procedure: inferior alveolar nerve lateralization and dental implant placement.; Procedure: platelet rich fibrin membrane around the nerve
- Group II (Active Comparator): inferior alveolar nerve lateralization for dental implant placement without placement of platelet rich fibrin membrane around the nerve.
  Interventions: Procedure: inferior alveolar nerve lateralization and dental implant placement.

INTERVENTIONS:
Procedure: inferior alveolar nerve lateralization and dental implant placement. — inferior alveolar nerve lateralization for placement of sufficiently long dental implants.
Procedure: platelet rich fibrin membrane around the nerve — platelet rich fibrin membrane is prepared from the patient's blood and placed around the nerve.
  Arms: Group I

SUMMARY:
In many cases the bone of the edentulous posterior mandibular regions is atrophied such that sufficiently long fixtures cannot be placed without encroaching on the inferior alveolar nerve so rehabilitation of these regions with severe ridge atrophy represents anatomical, surgical, and biological difficulties, and provides a challenge to the dental surgeon.

Several surgical techniques have been employed in an attempt to allow implant placement in these regions. one of these techniques is inferior alveolar nerve transposition or lateralization.

The lateralization of the inferior alveolar nerve has the advantages of that it allow placement of longer implants which gives better stability,but this technique has the disadvantage of high risk of temporary or permanent inferior alveolar nerve dysfunction.

In most of the cases of inferior alveolar nerve lateralization it is directly repositioned on the implant surface or a bone graft is placed in between them.

In a previous study on dogs found that presence of a resorbable membrane between the inferior alveolar nerve and the implant surface lead to the formation of a soft tissue zone between them while in the group where no membrane was used there was intimate contact between them.This intimate contact may lead to the dysfunction symptoms,also the intimate contact between the implant threads and the nerve act as a source of chronic irritation.

Platelet rich fibrin membrane is a platelet concentrate which allow slow and sustained release of high quantities of growth factors over long period of time thus improves healing of hard and soft tissue and optimizing wound healing.

in this study we will assess the effect of platelet rich fibrin membrane on the improvement of the neurosensory disturbances which occur after inferior alveolar nerve lateralization which considered as the main disadvantage of this technique.

DETAILED DESCRIPTION:
Background and rational:

In many cases the bone of the edentulous posterior mandibular regions is atrophied such that sufficiently long fixtures cannot be placed without encroaching on the inferior alveolar nerve so rehabilitation of these regions with severe ridge atrophy represents anatomical, surgical, and biological difficulties, and provides a challenge to the dental team.

Several surgical techniques have been employed in an attempt to allow implant placement in these regions. These include bone grafting, distraction osteogenesis, inferior alveolar nerve transposition or lateralization (IANL), and placement of fixtures in a lingual position to the neurovascular bundle.

The lateralization of the inferior alveolar nerve(IAN) has the advantages of that it allow placement of longer implants, gives better initial stability due to bicortical anchorage, and reduces the treatment time. Also it increases the resistance to the occlusal forces and improves the proportion between the implant and prosthesis.

This technique has the disadvantage of it is a complex procedure, with a high risk of complications which include temporary or permanent inferior alveolar nerve dysfunction.

In most of the cases of inferior alveolar nerve lateralization it is directly repositioned on the implant surface or a bone graft is placed in between them.

In a previous study on dogs it was found that presence of a resorbable membrane between the inferior alveolar nerve and the implant surface lead to the formation of a soft tissue zone between them (average distance was 348.3µm) while in the group where no membrane was used there was intimate contact between them (average distance was 39.8µm).This intimate contact may lead to the dysfunction symptoms or at least it does not prevent thermal conduction via implant surface,also the intimate contact between the implant threads and the nerve act as a source of chronic irritation which could induce longstanding edema and formation of intraneural fibrotic scar.

Platelet rich fibrin membrane is a second generation of platelet. It consist of high concentrate of collected platelets which allow slow and sustained release of high quantities of growth factors such as (Transforming Growth Factor b-1 (TGFbeta-1), platelet derived growth factor; vascular endothelial growth factor( VEGF) and an important coagulation matricellular glycoprotein wish is thrombospondin-1(TSP-1) over long period of time thus improves healing of hard and soft tissue and optimizing wound healing.

In addition it has advantage over other resorbable membranes because they are entirely autologous, simple in preparation method and low in cost.

In a previous study on rats the effect of platelet rich fibrin on sciatic nerve injury was studied, excision of 10 mm of the sciatic nerve was done then the nerve was bridged with a silicon tube filled with fragments of platelet rich fibrin. The walking track test showed significant improvement of functional recovery in the platelet rich fibrin group.

In the current literature there were no Randomized Clinical Trials (RCTs) that have evaluated the effect of platelet rich fibrin membrane on the neurosensory function of the inferior alveolar nerve after its lateralization and prevention of nerve dysfunction, so in this study we will assess the effect of platelet rich fibrin membrane on the improvement of the neurosensory disturbances which occur after inferior alveolar nerve lateralization and considered the main disadvantage of this technique.

Objectives of the study:

Assessment of the effect of platelet rich fibrin membrane on improvement of neurosensory disturbance of the inferior alveolar nerve after its lateralization. This assessment will be performed through:

A) Subjective assessment:

Using visual analogue scale.

b) Clinical assessment: using three tests:

1. Static light touch detection test.
2. Brush stroke discrimination test.
3. Tactile discrimination test.

   c) electrophysiological assessment: electro somatosensory evoked potential test of the inferior alveolar nerve.

   Study setting:

   Study is to be conducted on patients attending outpatient clinic in academic hospital of Faculty of Oral and Dental Medicine Cairo University department of oral and maxillofacial surgery, Egypt the Oral and Maxillofacial Surgery Department - Cairo University, Egypt.

   Diagnostic procedures:
   * all Patients with unilateral or bilateral posterior atrophic mandible (vertical defect) will undergo radiographic examination using cone beam computed tomography.
   * The side of the mandible (right or left) which has insufficient bone height above the inferior alveolar canal less than 8mm will be included in the study.
   * Participants will be given a brief explanation about the surgery and they were informed about possible alterations in lip sensation; any questions were fully answered and the patients will sign informed consents prior to the surgery.
   * Eligible sides will be randomized in equal proportions between two groups; Group I (study group) platelet rich fibrin group and Group II (control group).

   Criteria for discontinuing or modifying intervention:

   No protocol for discontinuation of the procedure as any complication occurs will be recorded and managed.

   Strategies to improve adherence to intervention. Face to face adherence reminder session will take place to stress on the importance of the follow up and post-operative instructions.

   The patient is informed with the importance of the follow up period until final loading of the implants after 6 months.

   Recruitment strategy:
   * Patients fulfilling the inclusion criteria and signed the informed consent will be selected from the outpatient clinic of the Oral and Maxillofacial Surgery Department - Cairo University
   * Screening of patients will continue until the target population is achieved

   Randomization method and allocation concealment mechanism:

   All patients who give consent for participation and who fulfill the inclusion criteria will be randomized.

   Sequence generation:

   Enrolled patients will be randomly distributed between the two groups (12 side in two categories) using online randomization program: http://www.Random.org.

   Allocation concealment:

   The numbers from 1 to 12 will be written in an eight folded papers each one will be placed in an opaque sealed envelope.

   participant with one side (right or left) included in the study will choose one of these envelopes which will determine the participant group according to the table obtained from random.org.while the participant with two sides (right and left) included in the study will choose two envelopes, the first envelope is for the right side and the second one is for the left side.

   The allocation key will be only with the study supervisor.

   Blinding:

   Patient and data analyst blinded.

   Data collection, management and analysis:

   Plans to promote participant retention and complete follow- up
   * Telephone numbers of all patients included the study will be recorded as a part of the written consent.
   * All patients will be given a phone call at the time of the pre-determined follow up dates.
   * These calls will be the responsibility of the assessor.

   Data management:
   * All data will be entered electronically.
   * Patient files are to be stored in numerical order and stored in secure and accessible place.

   Harms:

   Any possible adverse effects of the intervention will be recorded, documented and managed.

   Protocol amendments:

   Any modifications to the protocol which may impact on the conduct of the study, potential benefit of the patient or may affect patient safety, including changes of study objectives, study design, sample sizes, study procedures, or significant administrative aspects will require a formal amendment to the protocol. Such amendment will be agreed upon by the Council of oral and maxillofacial surgery department.

   Consent:

   Researcher will discuss the trial with all patients. Patients will then be able to have an informed discussion with the researcher. Researcher will obtain written consent from patients willing to participate in the trial. All consent forms will be in Arabic language.

   Confidentiality:

   All study-related information will be stored securely. All participant information will be stored in locked file cabinets in areas with limited access. Reports, data collection, process, and administrative forms will be identified by a coded identification number (ID) only to maintain participant confidentiality. All records that contain names or other personal identifiers will be stored separately from study records identified by code number. All local databases will be secured with password protected access systems.

   Access to data:

   All Principal Investigators will be given access to the data sets. All data sets will be protected by password. To ensure confidentiality, data dispersed to project team members will be blinded of any identifying participant information.

   Ancillary and post-trial care:

   All patients will be followed up until patients' satisfactions occur.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring dental implants placement in the posterior region and has insufficient bone height above the inferior alveolar canal to accommodate for implant placement.
* Patients should be free from any systemic conditions that may affect normal healing.

Exclusion Criteria:

* Patients with systematic disease that may complicate healing.
* Uncontrolled diabetic patient.
* Patients with advanced osteoporosis.
* Patients under bisphosphonates treatment.
* Heavy smoker patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Subjective assessment of the change in the neurosensory function of inferior alveolar nerve | pre-operative assessment (base line) and 1 week,2 weeks, 1 month, three months,six months postoperative
  a 10 cm, 5 degree visual analogue scale with divisions at 2.5 cm intervals, the divisions on the VAS was:
  1. Complete absence of sensations.
  2. Almost no sensation.
  3. Reduced sensation.
  4. Almost normal sensation.
  5. Fully normal sensation. Patients were asked to mark "x" on the line at each testing session that represent their opinion about sensation of the lower lip.

SECONDARY OUTCOMES:
clinical assessment of the change in the neurosensory function of inferior alveolar nerve: | pre-operative assessment (base line) and 1 week,2 weeks, 1 month, three months,six months postoperative.
  Static light touch detection test:
  using the von-Frey technique with the Semmes-Weinstein monofilaments, a series of nylon monofilaments of varying thickness that exert different pressures when pressed against the skin.
  the patient closes his eyes and says "yes" or "no" response if he feels a light touch, the patient should respond to two of three correct as an appropriate response. If not, the process should be repeated with increasingly stiffer monofilaments.
clinical assessment of the change in the neurosensory function of inferior alveolar nerve : | pre-operative assessment and (base line) 1 week,2 weeks, 1 month, three months,six months postoperative.
  Brush stroke discrimination test:
  the brush is rubbed across the tested area in anterior or posterior direction and the patient will give negative or positive response and determine the direction of the stroke.
clinical assessment of the change in the neurosensory function of inferior alveolar nerve | pre-operative assessment (base line) and 1 week,2 weeks, 1 month, three months,six months postoperative.
  Tactile discrimination test (two point discrimination test) the two points of the caliper are opened progressively in 1 mm increments until the patient can discriminate two points of contact at which the distance between the two points is recorded.

OTHER OUTCOMES:
electrophysiological assessment of the change in the neurosensory function of the inferior alveolar nerve | pre-operative assessment (base line) and two weeks postoperative
  electro-somatosensory evoked potential test of the inferior alveolar nerve ,the test will be performed in the neurophysiology unit ,cairo university the latency and amplitude of each evoked potential are measured

CONTACTS AND LOCATIONS:
Overall Officials: Eman S Shalaby, ass.lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry ,Cairo university, Cairo, Egypt